CLINICAL TRIAL: NCT03639389
Title: Randomised Comparison Between Spinal/GA or GA Alone Following Robot-assisted Laparoscopic Prostatectomy. Stress Response, Pain, Recovery and Home Discharge
Brief Title: Postoperative Pain, Recovery and Discharge Following Robot-assisted Laparoscopic Prostatectomy
Acronym: RAPID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-06
Record Dates: First submitted 2018-08-06; First posted 2018-08-21 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Radical Prostatectomy; Postoperative Pain
Keywords: Robot assisted surgery; Prostatectomy; Spinal anesthesia; Postoperative pain; Home discharge
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Analgesics; Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Morphine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, observer-blinded
Who Masked: Outcomes Assessor
Masking Description: Outcome observer blinded to method of analgesia (spinal/no-spinal)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesics, multimodal (Active Comparator): Combination of paracetamol, non-steroidal anti-inflammatory drug and morphine as analgesics
  Interventions: Drug: Analgesics
- Bupivacaine (Experimental): Spinal anesthetic with bupivacain + fentanyl/sufentanil
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Spinal anesthesia with a combination of bupivacaine and fentanyl or sufentanil
  Other Names: Marcain spinal
  Arms: Bupivacaine
Drug: Analgesics — Combination of paracetamol + non-steroidal anti-inflammatory drug + morphine to all patients
  Other Names: paracetamol + NSAID + morphine
  Arms: Analgesics, multimodal

SUMMARY:
Prostate cancer is the commonest cancer form in men in Northern Europe. Management of the cancer often includes surgical removal of the primary tumor. In the last 5-10 years, robot assisted laparoscopic prostatectomy (RALP) has become common. Good pain relief is central to early mobilization and greater patient satisfaction. Randomized controlled studies on pain relief following RALP are few and the role of spinal analgesia in pain management following robotic surgery has not been described. Techniques available for pain relief following RALP include spinal anesthesia with or without opiates, intravenous analgesia with morphine or a multimodal pain management technique using a combination of several analgesics. Spinal anesthesia and analgesia reduces the surgical stress and inflammatory response following laparoscopic colorectal surgery and may offer similar benefit even during RALP.

Early perioperative complications may cause postoperative morbidity following robotic surgery, and sometimes delay home discharge. Since all robotic operations in the pelvic region are performed in a deep Trendelenberg position, this can even have negative consequences for the heart, brain and the lungs. Cardiac complications in the form of minimal cardiac injury or mild heart failure have not been previously studied following RALP. Additionally, patients are sometimes delirious in the early postoperative period following RALP. The precise cause for this remains unclear and may be related to pain, cognitive dysfunction or an urge to pass urine despite a urinary catheter.

In addition to good postoperative pain relief, early postoperative mobilization and home discharge are important milestones in recovery of full function following major surgery. With improvement in surgical technique, the time has come to evaluate if RALP can be performed on an ambulatory basis. The main aims of this study are:

1. Can RALP be performed on an ambulatory basis and patients ready to be discharged home at 8 pm?
2. To determine if spinal anesthesia reduces pre-discharge pain intensity, stress response and other perioperative side effects.
3. Is sufentanil or fentanyl the analgesic of choice when administered spinally together with bupivacaine as an analgesic.
4. To determine the frequency and severity of cardiac and respiratory complications in the steep Trendelenberg position during RALP.
5. To assess the quality of recovery, quality of life and activities of daily living following ambulatory RALP?

DETAILED DESCRIPTION:
Prospective, randomized study blinded to observers (spinal or no-spinal). All formal approvals will be obtained from different authorities prior to study start. It will be registered in an international database (clinicaltrials.gov).

Patients > 18 years, ASA I-III, undergoing RALP will be included into the study. Patients on chronic opiate medication, those with contraindications to spinal anesthesia or allergy to any component drugs used during spinal anesthesia or other analgesics used in the study will be excluded. Patients living alone or having no adult at home to look after them during the first 24 h after home discharge will also be excluded. Informed written consent will be obtained from all patients. On the morning of surgery, all patients will receive paracetamol 1 g orally 1 h before planned surgery, and will be randomized to one of two groups as shown below:

Robot-assisted laparoscopic prostatectomy (RALP) (morning surgery)

1. Group MM: This group of patients will not receive spinal anesthesia but have multimodal pain management including COX-2 blockers, pregabalin and oxycontin for pain management
2. Group SF (Spinal/Fentanyl): Spinal anesthesia with bupivacaine 12.5 mg+fentanyl 15 ug Robot-assisted laparoscopic prostatectomy (RALP) (afternoon surgery)

1. Group MM: This group of patients will not receive spinal anesthesia but have multimodal pain management including COX-2 blockers, pregabalin and oxycontin for pain management 2. Group SS (Spinal/Sufentanil): Spinal anesthesia with bupivacaine 12.5 mg+sufentanil 5 ug

Anesthesia will be standardized in all other aspects in all groups and basically include propofol for induction, rocuronium as muscle relaxant, sevoflurane and remifentanil for pain management and betamethasone + ondansetron as prophylaxis against post-operative nausea or vomiting (PONV). Surgery will also be standardized in all patients and follow the routines already established in the hospital.

At the end of surgery, patients will be transferred to the post-anesthesia care unit (PACU) where they will remain for 4 h observation and subsequently transferred to the general surgical wards for observation and discharge home. All measurement times will be taken from the end of surgery, which will be considered as t = 0.

The following parameters will be recorded:

1. Total morphine consumption during 0-4, 4-home discharge and analgesic supplements after home discharge and up to 1 week will be recorded. Time to first morphine administration after surgery will be registered.
2. Blood tests for measurement of cortisol, glucose, insulin, creatinine, NTproBNP and hsTnT will be taken at fixed time points before and after surgery.
3. Pain intensity will be registered using NRS after 1, 2, 3, 4 and every 4 h until home discharge, and thereafter every 24 h for 1 week.
4. All side effects (PONV, pruritus, respiratory depression, oxygen saturation and need for supplementary oxygen) and complications (bleeding, reoperation, pneumothorax etc.) will be recorded. Postoperative delirium will be assessed 0-2 h postoperatively. Prolonged PACU stay or re-admission to PACU will be registered. Clavien-Dindo classification for grade of complication will be registered as also Postoperative Morbidity score (POMS).
5. Respiratory function will be recorded in the following ways: blood gas (after 1 and 4 h), saturation, spirometry, maximum expiratory pressure preoperatively and after 4 h. Need for supplementary oxygen to maintain SpO2 > 93% will be registered.
6. Time to mobilization, time to discharge to the general ward (from PACU), "home readiness" (primary endpoint) and home discharge will be registered in accordance with standardized criteria. Criteria for home readiness: normal vital signs, pain intensity < 4 (NRS 0-10), minimal or no postoperative nausea or vomiting, able to sit, walk and go unhindered, no surgical complication (bleeding, fever), fully awake and able to follow instructions (normal cognition), normally functioning urinary catheter and an adult at home during the first 24 h after discharge home).
7. Quality of Recovery 15 (QoR 24) will be measured before home-discharge and after 24 h using a standardized questionnaire.
8. Quality of life will be measured preoperatively and after 7 and 30 days using the questionnaire EQ5D and WHODAS.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Elective robot-assisted laparoscopic prostatectomy Karolinska Hospital

Exclusion Criteria:

* Communication limitations (language, mental)
* Chronic opiate use
* Allergy to NSAID
* Coagulation problems preventing administration of spinal analgesia

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males undergo this procedure
Enrollment: 211 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Number of patients ready for home discharge at 8 pm after surgery | With 12 h of surgery start
  Number of patients ready to be discharged home after surgery when using a standardized home-discharge criteria

SECONDARY OUTCOMES:
Pain intensity | 7 days postoperatively
  Intensity of pain recorded using numeric rating score at defined time intervals postoperatively
Stress markers in plasma | 24 hours
  Blood glucose, cortisol and insulin
Quality of Recovery | 3 days postoperatively
  Quality of recovery will be measured at defined time intervals using a standardized questionnaire
Quality of life after surgery | 30 days postoperatively
  Quality of life will be measured at defined time intervals pre- and postoperatively using a standardized questionnaire
Amount (mg) of morphine administered as rescue analgesic at 12 and at 24 h | At 12 hours and 24 hours postoperatively
  Total amount of rescue analgesics (morphine) administered to achieve good analgesia and mild pain (NRS < 4)

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Björne, MD, PhD, Study Director — Karolinska Hospital
Locations (2):
- Sweden (2):
  - Karolinska Hospital, Solna, Stockholm
  - Capio St Görans Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
Not known currently